CLINICAL TRIAL: NCT01332071
Title: Assessment of Relative Bioavailability of Avandamet 4 mg + 1000 mg (GSK) in the Form of Film Coated Tablets Versus Avandamet 2 mg + 500 mg (GSK) in the Form of Film Coated Tablets, in Healthy Volunteers After Feeding Standardized, Using Liquid Chromatography.
Brief Title: Avandamet Bioequivalence Study Brazil - Fed Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 114040
Record Dates: First submitted 2010-08-31; First posted 2011-04-08 (Estimated); Results first posted 2011-04-08 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Metformin; Rosiglitazone; Healthy volunteers; Avandamet; Fed conditions; Bioequivalence
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Avandamet test product (Active Comparator): Test product: Avandamet (Rosiglitazone Maleate + Metformin) 4 miligrams (mg) + 1000 mg in Period 1, followed by a 7-day washout period during which no medication was administered, followed by reference product: Avandamet (Rosiglitazone Maleate + Metformin) 2 mg + 500 mg in Period 2
  Interventions: Drug: Rosiglitazone Maleate + Metformin 4 miligrams (mg) + 1000 mg
- Avandamet reference product (Active Comparator): Reference product: Avandamet (Rosiglitazone Maleate + Metformin) 2 miligrams (mg) + 500 mg in Period 1; followed by a 7-day washout period during which no medication was administered; followed by test product: Avandamet (Rosiglitazone Maleate + Metformin) 4 mg + 1000 mg in Period 2
  Interventions: Drug: Rosiglitazone Maleate + Metformin 2 miligrams (mg) + 500 mg

INTERVENTIONS:
Drug: Rosiglitazone Maleate + Metformin 2 miligrams (mg) + 500 mg — Avandamet reference product
  Arms: Avandamet reference product
Drug: Rosiglitazone Maleate + Metformin 4 miligrams (mg) + 1000 mg — Avandamet test product
  Arms: Avandamet test product

SUMMARY:
The study is prospective, open-label, randomized, crossover, with 02 treatments, 02 sequences, and 02 periods. The volunteers received, in each period, the reference or the test formulation after standardized meals.

DETAILED DESCRIPTION:
This is an open-label, randomized, crossover study with 02 treatments, 02 sequences, and 02 periods, in which the healthy volunteers received, in each period, the test or the reference formulation after standardized meals. Test product is Rosiglitazone Maleate + Metformin - Avandamet 4 mg + 1000 mg (GlaxoSmithKline Brasil Ltda) in the form of film coated tablets. Reference product is Rosiglitazone Maleate + Metformin - Avandamet 2 mg + 500 mg (Glaxo Smith Kline Brasil Ltda) in the form of film coated tablets. The population is composed by 26 healthy volunteers, adults, of both genders and their ages varied between 18 and 50 years. Their body mass index (BMI) varied between 18,5 and 25. There are no restrictions regarding the ethnic group. The relative bioavailability of the two formulations, after oral administration, will be evaluated based on statistical comparisons of relevant pharmacokinetic parameters obtained from data of drug concentration in blood.

ELIGIBILITY:
EXCLUSION CRITERIA:

* The volunteer has a known hypersensitivity to the study drug or to compounds chemically related;
* History or presence of hepatic or gastrointestinal illnesses, or other condition that interferes over the drug's absorption, distribution, excretion or metabolism;
* History of neurological, endocrine, pulmonary, hamatologic, immune, brain, metabolic or cardiovascular illness;
* Hypo or hypertension of any etiologic that needs pharmacologic treatment;
* The results of the laboratory exams are out of the values considered as normal according this protocol's rules, unless that they are considered as clinically irrelevant by the investigator;
* Has history of alcohol or drugs abuse;
* History of use drug inducing and/or inhibitors of hepatic metabolism within 30 days prior to drug study administration;
* Use of MAO inhibitors two weeks before the start of treatment; - Use of inhibitors of 5-TH reuptake,
* Pregnancy or breastfeeding,
* Smoking;
* Use of regular medication within 4 weeks prior to study iniciation;
* Use of experimental drug or participation in any clinical study within 6 months prior to study iniciation.

INCLUSION CRITERIA:

* Age between 18 and 50 years;
* Body mass index ≥ 18,5 and ≤25,0, can vary up to 15% for the upper limit (18,5 to 28,75);
* Good health conditions;
* Obtain the Informed Consent's signed.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2009-11-24 (Actual); Primary Completion 2009-12-06 (Actual); Study Completion 2009-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Goiânia, Goiás, Brazil

REFERENCES:
- See also: Results for study 114040 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114040?search=study&search_terms=114040#rs

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Product in Period 1; Reference Product in Period 2: Test product: Rosiglitazone Maleate + Metformin film coated tablets (Avandamet) 4 milligrams (mg) + 1000 mg (GlaxoSmithKline Brasil Ltda) in Period 1; followed by a 7-day washout period during which no medication was administered; followed by reference product: Avandamet 2 mg + 500 mg (GlaxoSmithKline Brasil Ltda) in Period 2
- Reference Product in Period 1; Test Product in Period 2: Reference product: Avandamet 2 mg + 500 mg in Period 1; followed by a 7-day washout period during which no medication was administered; followed by test product: Avandamet 4 mg + 1000 mg in Period 2
Period: Period 1
Arm/Group | Test Product in Period 1; Reference Product in Period 2 | Reference Product in Period 1; Test Product in Period 2
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0
Period: 7-Day Washout Period
Arm/Group | Test Product in Period 1; Reference Product in Period 2 | Reference Product in Period 1; Test Product in Period 2
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Test Product in Period 1; Reference Product in Period 2 | Reference Product in Period 1; Test Product in Period 2
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Participants Receiving Both Test and Reference Product: Participants receiving either test product: Avandamet 4 mg + 1000 mg in Period 1; followed by reference product: Avandamet 2 mg + 500 mg in Period 2 or reference product in Period 1 and test product in Period 2
Arm/Group | Participants Receiving Both Test and Reference Product
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.77 (6.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: AUC0-t of Rosiglitazone Maleate
Description: The area under the plot of plasma concentration of drug against time after drug administration is defined as the area under the curve (AUC). The AUC 0-t is calculated from time 0 (prior to administration of medication) to time t (the time of the last quantifiable concentration). The AUC is of particular use in estimating the bioavailability of drugs, by measuring the extent of absorption. ng, nanograms; ml, milliliter.
Time Frame: Day 1 (day that blood collection started) and Day 2 (Period 1) and Days 8 and 9 (Period 2)
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: ng per hour per ml (ng.h/ml)
Groups:
- Test Product: Test product: Rosiglitazone Maleate 4 mg in both periods
- Reference Product: Reference product: Rosiglitazone Maleate 2 mg in both periods
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 26 | 26
ng per hour per ml (ng.h/ml) | 1731.22 (510.47) | 1770.93 (469.14)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — This is a bioequivalence study. The study was performed to fulfill a specific regulatory demand of the Brazilian Regulatory Agency - ANVISA, in order to register a new dosage of medication; Ratio T formulation/R formulation = 96.58, 90% CI 2-sided [93.44 to 99.83] — The ratio between the geometric means of the test (T) and reference (R) formulations was calculated

2. Primary Outcome: Cmax of Rosiglitazone Maleate
Description: Cmax is defined as the maximum or "peak" concentration of a drug observed after its administration. Cmax is one of the parameters of particular use in estimating the bioavailability of drugs, by measuring the total amount of drug absorbed.
Time Frame: Day 1 (day that blood collection started) and Day 2 (Period 1) and Days 8 and 9 (Period 2)
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 26 | 26
ng/ml | 265.45 (44.33) | 270.97 (48.32)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio T formulation/R formulation = 97.76, 90% CI 2-sided [93.25 to 102.50] — The ratios between the geometric means of the test (T) and reference (R) formulations was calculated

3. Primary Outcome: AUC0-infinity of Rosiglitazone Maleate
Description: The area under the plot of plasma concentration of drug against time after drug administration is defined as the area under the curve (AUC). The AUC0-infinity is calculated from time 0 (prior to administration of medication) to infinity (the time of complete elimination of the drug). The AUC is of particular use in estimating the bioavailability of drugs, by measuring the extent of absorption.
Time Frame: Day 1 (day that blood collection started) and Day 2 (Period 1) and Days 8 and 9 (Period 2)
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: ng.h/ml
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 26 | 26
ng.h/ml | 1776.28 (519.63) | 1825.35 (494.35)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio T formulation/R formulation = 96.47, 90% CI 2-sided [93.32 to 99.72] — The ratio between the geometric means of the test (T) and reference (R) formulations was calculated

4. Primary Outcome: AUC0-t of Metformin Hydrochloride
Description: The area under the plot of plasma concentration of drug against time after drug administration is defined as the area under the curve (AUC). The AUC0-t is calculated from time 0 (prior to administration of medication) to time t (the time of the last quantifiable concentration). The AUC is of particular use in estimating the bioavailability of drugs, by measuring the extent of absorption. ng, nanograms; ml, milliliter.
Time Frame: Day 1 (day that blood collection started) and Day 2 (Period 1) and Days 8 and 9 (Period 2)
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: ng.h/ml
Groups:
- Test Product: Test product: Metformin Hydrochloride 1000 mg in both periods
- Reference Product: Reference product: Metformin Hydrochloride 500 mg in both periods
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 26 | 26
ng.h/ml | 9623.4 (2175.4) | 10074.4 (2411.7)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio T formulation/R formulation = 95.79, 90% CI 2-sided [91.67 to 100.10] — The ratios between the geometric means of the test (T) and reference (R) formulations was calculated

5. Primary Outcome: AUC0-infinity of Metformin Hydrochloride
Description: as for outcome 3
Time Frame: Day 1 (day that blood collection started) and Day 2 (Period 1) and Days 8 and 9 (Period 2)
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: ng.h/ml
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 26 | 26
ng.h/ml | 10419.8 (2198.2) | 11063.7 (2798.3)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio T formulation/R formulation = 94.86, 90% CI 2-sided [90.70 to 99.22] — The ratios between the geometric means of the test (T) and reference (R) formulations was calculated

6. Primary Outcome: Cmax of Metformin Hydrochloride
Description: as for outcome 2
Time Frame: Day 1 (day that blood collection started) and Day 2 (Period 1) and Days 8 and 9 (Period 2)
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 26 | 26
ng/ml | 1623.6 (326.5) | 1663.9 (370.2)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio T formulation/R formulation = 97.88, 90% CI 2-sided [93.15 to 102.86] — The ratios between the geometric means of the test (T) and reference (R) formulations was calculated

ADVERSE EVENTS:
Arm/Group | Test Product in Period 1; Reference Product in Period 2 | Reference Product in Period 1; Test Product in Period 2
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 13/13 | 13/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Product in Period 1; Reference Product in Period 2 (N=13) | Reference Product in Period 1; Test Product in Period 2 (N=13)
Cephalea (General disorders) | 3 | 0
Tension cephalea (General disorders) | 1 | 0
Frontal cephalea (General disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 3
Diarrhea with semi liquid stool (Gastrointestinal disorders) | 1 | 1
Evacuation of liquid stool (Gastrointestinal disorders) | 1 | 0
Post-study increased urea (Renal and urinary disorders) | 1 | 0
Post-study altered urine exam (Renal and urinary disorders) | 12 | 8
Post-study increased leucocytes (Blood and lymphatic system disorders) | 1 | 1
Post-study increased total cholesterol (Blood and lymphatic system disorders) | 0 | 1
Post-study increased triglycerides (Blood and lymphatic system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.